CLINICAL TRIAL: NCT03572582
Title: A Phase II Single-arm, Open-label Study of Transarterial Chemoembolization (TACE) in Combination With Nivolumab Performed for Intermediate Stage Hepatocellular Carcinoma (HCC)
Brief Title: Transarterial Chemoembolization in Combination With Nivolumab Performed for Intermediate Stage Hepatocellular Carcinoma
Acronym: IMMUTACE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIO-Studien-gGmbH (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AIO-HEP-0217; 2017-003553-42 (EudraCT Number); CA209-9KK (Other Grant/Funding Number: Bristol-Myers Squibb)
Record Dates: First submitted 2018-05-29; First posted 2018-06-28 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: Carcinoma, Hepatocellular; Hepatic Carcinoma; Hepatocellular Cancer
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TACE in combination with nivolumab (Experimental): Treatment will be divided into 4-week cycles from the starting date of TACE. The second TACE will be repeated on day 1 (± 4 days) of cycle 3 (after 8 weeks ± 4 days). Nivolumab will be initiated on day 2-3 after the first TACE session. Nivolumab will be administered every two weeks (240mg fixed dose IV) until disease progression for up to two years.
  Interventions: Drug: Nivolumab; Drug: TACE

INTERVENTIONS:
Drug: Nivolumab — Nivolumab therapy combined with standard TACE treatment
Drug: TACE — TACE is performed by using drug eluting beads

SUMMARY:
The IMMUTACE study evaluates the safety and the efficacy of the anti-programmed-death-1 antibody (anti-PD-1) nivolumab in combination with transarterial chemoembolization (TACE) in patients with multinodular, intermediate stage hepatocellular carcinoma (HCC) as first line therapy.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is one of the most lethal and prevalent cancers worldwide. The prognosis of patients with HCC is dismal and the mortality rates are almost the same as the incidence rates.

The transarterial chemoembolization (TACE) is commonly used to act locally in the intermediate disease stage and is the most common first-line treatment in patients with HCC. Early randomized trials and more recent reviews and meta-analyses reported improved survival rates of patients with unresectable lesions managed with TACE so that TACE has been accepted as the standard treatment for intermediate stage disease. However, outcome of patients treated with TACE in real-life cohorts is still very poor with median overall survival (OS) of 20 months or less.

In order to increase the outcome of TACE, several trials have analyzed the combination of TACE with sorafenib and other anti-angiogenic agents. However, none of the trials have reported an improved overall survival for patients treated with the combination of TACE and sorafenib. Early clinical data already support a safe combination of immune checkpoint inhibition with TACE. Moreover, preliminary data from the CheckMate-040 trial strongly suggest that nivolumab has clinical activity and is tolerable in patients with HCC, including those with hepatitis B or hepatitis C virus (HCV) infection.

Therefore, the aim of this study is to evaluate the safety and efficacy of TACE in combination with nivolumab in patients with intermediate stage HCC.

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent including participation in translational research and any locally-required authorization (EU Data Privacy Directive in the EU) obtained from the subject prior to performing any protocol-related procedures, including screening evaluations.
2. Age ≥ 18 years at time of study entry
3. Multinodular or large, solitary HCC, not eligible for resection or local ablation, Tumor burden below 50% of liver volume.
4. Histologically confirmed diagnosis of HCC.
5. At least one measurable site of disease as defined by modified RECIST (mRECIST) criteria with spiral CT scan or MRI.
6. Child-Pugh A, performance status (PS) ≤ 2 (ECOG scale).
7. Subjects with chronic HBV infection must have HBV DNA viral load < 100 IU/mL at screening. In addition, they must be on antiviral therapy per regional standard of care guidelines prior to initiation of study therapy.
8. Life expectancy of at least 12 weeks.
9. Adequate blood count, liver-enzymes, and renal function: Haemoglobin ≥ 8.5 g/dL, absolute neutrophil count ≥ 1,500/L, platelets ≥70 x103/L; Total bilirubin ≤ 3x upper normal limit; Aspartate Aminotransferase (SGOT), Alanine aminotransferase (SGPT) ≤ 5 x upper normal limit (ULN); International normalized ratio (INR) ≤1.25; Albumin ≥ 31 g/dL; Serum Creatinine ≤ 1.5 x institutional ULN or creatinine clearance (CrCl) ≥ 30 mL/min (if using the Cockcroft-Gault formula )
10. Female patients with reproductive potential must have a negative urine or serum pregnancy test within 7 days prior to start of trial.
11. Subject is willing and able to comply with the protocol for the duration of the study including undergoing treatment, adherence to contraceptive measures, scheduled visits and examinations including follow up.

Exclusion criteria:

Methodological or clinical criteria:

1. Diffuse HCC or presence of vascular invasion or extrahepatic spread with the following exceptions:

   1. Invasion of a segmental portal vein or hepatic veins
   2. Limited extrahepatic metastases with one organ system manifestations, e.g. lymphnodal, pulmonary, ossary metastases. For lymphnodal metastases Maximum three metastases, maximum 2 cm in the longest diameter, and for all other metastases only solitary metastases, maximum 2 cm in the longest diameter, are allowed.
2. Patients on a liver transplantation list or with advanced liver disease as defined below:

   1. Encephalopathy;
   2. Untreatable ascites.
3. Any contraindications for hepatic embolization procedures:

   1. Known hepatofugal blood flow;
   2. Known porto-systemic shunt;
   3. Impaired clotting test (platelet count <70 x103/L, INR >1.25);
   4. Renal failure/ insufficiency requiring hemo-or peritoneal dialysis;
   5. Known severe atheromatosis;
   6. Total thrombosis or total invasion of the main branch of the portal vein.
4. History of cardiac disease:

   1. Congestive heart failure >New York Heart Association (NYHA) class 2;
   2. Active coronary artery disease (CAD) (myocardial infarction ≥ 6 months prior to study entry is allowed);
   3. Cardiac arrhythmias (>Grade 2 NCI-CTCAE Version 4.03) which are poorly controlled with anti-arrhythmic therapy or requiring pace maker;
   4. Uncontrolled hypertension;
   5. Clinically significant gastrointestinal bleeding within 4 weeks prior to start of study treatment (TACE + nivolumab)
5. Thrombotic or embolic events such as cerebrovascular accident (including transient ischemic attacks), deep vein thrombosis or pulmonary embolism within the 6 months Prior to the first dose of study drug with the exception of thrombosis of a segmental portal vein.
6. Prior systemic anti-cancer therapy OR endocrine- OR immunotherapy
7. Prior treatment with TACE
8. RFA and resection administered less then 4 weeks prior to study treatment start.
9. Radiotherapy administered less then 4 weeks prior to study treatment start.
10. Major surgery within 4 weeks of starting the study treatment OR subjects who have not recovered from effects of major surgery.
11. Patients with second primary cancer, except adequately treated basal skin cancer or carcinoma in-situ of the cervix.
12. Immunocompromised patients, e.g. patients who are known to be serologically positive for human immunodeficiency virus (HIV).
13. Participation in another clinical study with an investigational product during the last 30 days before inclusion or 7 half-lifes of previously used trial medication, whichever is longer.
14. Previous treatment in the present study (does not include screening failure).
15. Any condition or comorbidity that, in the opinion of the investigator, would interfere with evaluation of study Treatment or interpretation of patient safety or study results, including but not limited to:

    1. history of interstitial lung disease
    2. Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) coinfection (i.e double infection)
    3. known acute or chronic pancreatitis
    4. active tuberculosis
    5. any other active infection (viral, fungal or bacterial) requiring systemic therapy
    6. history of allogeneic tissue/solid organ transplant
    7. diagnosis of immunodeficiency or patient is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of nivolumab-monotherapy treatment.
    8. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Exceptions: Subjects with vitiligo, hypothyroidism, diabetes mellitus type I or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with Hashimoto thyroiditis, hypothyroidism stable on hormone replacement or psoriasis not requiring treatment are not excluded from the study.
    9. Live vaccine within 30 days prior to the first dose of nivolumab-monotherapy treatment or during study treatment.
    10. History or clinical evidence of Central Nervous System (CNS) metastases Exceptions are: Subjects who have completed local therapy and who meet both of the following criteria: I. are asymptomatic and II. have no requirement for steroids 6 weeks prior to start of nivolumab-monotherapy treatment. Screening with CNS imaging (CT or MRI) is required only if clinically indicated or if the subject has a history of CNS

    Drug related criteria:
16. Medication that is known to interfere with any of the agents applied in the trial.
17. Has known hypersensitivity to nivolumab or any of the constituents of the products.
18. Any other efficacious cancer treatment except protocol specified treatment at study start.
19. Patient has received any other investigational product within 28 days of study entry.
20. Prior therapy with an anti-Programmed cell death protein 1 (anti-PD-1), anti-PD-L1, anti-Programmed cell death-ligand 2 (anti-PD-L2), anti-CD137 (4-1BB ligand, a member of the Tumor Necrosis Factor Receptor (TNFR) family), or anti-Cytotoxic T-lymphocyte-associated antigen-4 (anti-CTLA-4) antibody (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).

    Safety criteria:
21. Female subjects who are pregnant, breast-feeding or male/female patients of reproductive potential who are not employing an effective method of birth control (failure rate of less than 1% per year). [Acceptable methods of contraception are: implants, injectable contraceptives, combined oral contraceptives, intrauterine pessars (only hormonal devices), sexual abstinence or vasectomy of the partner]. Women of childbearing potential must have a negative pregnancy test (serum β-HCG) at screening.

    Regulatory and ethical criteria:
22. Patient with any significant history of non-compliance to medical regimens or with inability to grant reliable informed consent.
23. Patient who has been incarcerated or involuntarily institutionalized by court order or by the authorities § 40 Abs. 1 S. 3 Nr. 4 Arzneimittelgesetz (AMG - German Drug Law).
24. Patients who are unable to consent because they do not understand the nature, significance and implications of the clinical trial and therefore cannot form a rational intention in the light of the facts [§ 40 Abs. 1 S. 3 Nr. 3a AMG].

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2018-06-14 (Actual); Primary Completion 2021-10-12 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Observation period max 42 months
  Objective Response Rate according to modified RECIST for HCC

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | max 42 months
  Progression according to mRECIST for HCC with the exception of new intrahepatic lesions, which are assessed to be treatable with one additional locoregional therapy. Progression following one additional locoregional treatment of such lesions according to mRECIST would be equivalent to failure of strategy.
Time to Progression (TTP) | max 42 months
  It is defined as the time from first TACE to the date of the first documented tumor progression according to the definition above.
Overall survival (OS) | max 42 months
  Overall survival is defined as the time from first TACE until death.
Duration of Response (OR) | max 42 months
  It is defined as time between the date of first radiographic documented objective response according to mRECIST for HCC and the date of the radiographic disease progression.
Objective Response Rate according to RECIST 1.1 | max 42 months
  A secondary objective is to estimate best ORR according to RECIST 1.1.
Time to Failure of Strategy (TTFS) | max 42 months
  Progression according to mRECIST for HCC with the exception of new intrahepatic lesions, which are assessed to be treatable with one additional locoregional therapy (TACE, radiofrequency ablation [RFA] / microwave ablation [MWA] or resection)
Quality of Life (QoL) | 36 moths
  EORTC-QLQ-C30 (European Organisation for Research and Treatment of Cancer - Quality of Life Core Questionnaire 30 items) Version 3.0. The QLQ-C30 is composed of multi-item scales and single-item measures, including five functional scales, three symptom scales, a global health Status / QoL scale, and six single items. All of the scales and single-item measures have a score range from 0 to 100. A high score shows a high response level. A high score for a functional scale represents a high / healthy level of functioning, a high score for the global health status / QoL represents a high QoL, but a high score for a symptom scale / item represents a high level of symptomatology / problems functional scales, three symptom scales, a global health status / QoL scale, and six single items.
Quality of Life (QoL) | 36 months
  EORTC-QLQ-HCC18 (European Organisation for Research and Treatment of Cancer - Quality of Life Core Questionnaire - Hepatocellular carcinoma module 18). The HCC18 module for patients with Hepatocellular carcinoma includes 18 items, conceptualised as consisting of 6 scales and 2 single items, which should always be complemented by the EORTC-QLQ-C30.
Incidence of Treatment Emergent Adverse Events as assessed by NCI CTCAE V4.03 (Safety and Tolerability) | 42 months
  Data will be obtained on vital signs, clinical parameters and feasibility of the regimen

CONTACTS AND LOCATIONS:
Overall Officials: Arndt Vogel, Prof.Dr., Principal Investigator — Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie & Endokrinologie
Locations (1):
- Medizinische Hochschule Hannover, Klinik für Gastroenterologie, Hepatologie & Endokrinologie, Hanover, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kloeckner R, Galle PR, Bruix J. Local and Regional Therapies for Hepatocellular Carcinoma. Hepatology. 2021 Jan;73 Suppl 1:137-149. doi: 10.1002/hep.31424. Epub 2020 Nov 6. No abstract available. PMID 32557715
- See also: Description AIO - Working Group for Medical Oncology from the German Cancer Society — http://www.aio-portal.de/
- See also: AIO-Studien-gGmbH — http://www.aio-studien-ggmbh.de/index.html